CLINICAL TRIAL: NCT02976805
Title: A Multi-centre Endoscopist Blinded Randomized Clinical Trial to Compare Two Bowel Preparations After a Colonoscopy With Inadequate Bowel Preparation
Brief Title: Multi-centre Failed Bowel Prep RCT
Acronym: B-CLEANR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other); Pendopharm (Industry); University of Alberta (Other); Université de Montréal (Other); McGill University (Other); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSREB108472
Record Dates: First submitted 2016-11-25; First posted 2016-11-29 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-01

CONDITIONS: Colonoscopy; Bowel Preparation
MeSH Terms: interventions — Bisacodyl; OOS-A regimen; Regimen B

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regimen A (Experimental): 4L PegLyte + 15 mg bisacodyl
  Interventions: Drug: 4L PegLyte + 15 mg bisacodyl
- Regimen B (Experimental): 6L PegLyte + 15 mg bisacodyl
  Interventions: Drug: 6L PegLyte + 15 mg bisacodyl

INTERVENTIONS:
Drug: 4L PegLyte + 15 mg bisacodyl — Randomized
  Other Names: Regimen A
  Arms: Regimen A
Drug: 6L PegLyte + 15 mg bisacodyl — Randomized
  Other Names: Regimen B
  Arms: Regimen B

SUMMARY:
This is a multi-centre randomized clinical trial comparing the efficacy of two different bowel preparation regimens for patients who have already failed a bowel preparation for colonoscopy.

DETAILED DESCRIPTION:
PURPOSE

The purpose of this multi-centre randomized clinical trial is to compare two bowel preparation regimens for patients who fail to cleanse their colon during their index colonoscopy. Although many clinical trials already exist examining the optimal bowel preparation for colonoscopy in general, surprisingly none address patients who failed bowel preparation in the past. Failure to achieve bowel preparation is a result of complex factors, including underlying colonic dysmotility, co-morbidities, and concurrent medication usage and is rarely the result of patient non-compliance.(1) Given the frequency of inadequate bowel preparation, its negative impact on colonoscopy quality, the increased risk for an adverse event, and the need to repeat the procedure, an important public health need exists to address this question urgently.(1) This study will use many of the same methodology and investigators as an ongoing Canadian multicenter study titled, "The Bowel CLEAnsing: a National initiative ( B-CLEAN) " but on a smaller scale to answer this question.

BACKGROUND

Adequate bowel preparation is a prerequisite for high quality colonoscopy and is needed to maximize visualization of the colonic mucosa.(1-4) Unfortunately, inadequate bowel preparation is common and reported to occur in 4% to 17% of cases.(5-12) Procedures with poor preparation are more likely to be incomplete, have an adverse event, and are less likely to detect polyps.(1, 9, 13) Repeat colonoscopies within one year have shown a 36% miss rate for advanced adenomas in these patients.(12) Recognizing the importance of high quality colonoscopy, Cancer Care Ontario and other provincial health authorities now track adequacy rates for bowel preparation.

In cases of poor bowel preparation, the colonoscopy must be repeated, exposing patients to another invasive procedure and adding additional costs to the healthcare system. Although health economic data regarding colonoscopy utilization in Canada is sparse, an illustrative example from the United States is possible. Assuming 14.2 million screening colonoscopies are performed annually in the United States (14) of which 5% have inadequate bowel preparation (6, 8), a total of 710,000 colonoscopies have to be repeated at a cost of $763 million dollars, based on a per case cost of $1,075.(15) This is likely an underestimation of the true cost due to exclusion of non-screening colonoscopies in the calculation and the use of a low colonoscopy cost estimate based on the Nationwide Colonoscopy Program for the Uninsured.(15)

There are numerous definitions of inadequate bowel preparation and the term's lack of specificity contributes to the varied incidence of inadequate bowel preparation reported in the literature. The Boston Bowel Preparation Scale (BBPS) is a user friendly validated measure that is based on three colonic segment scores (right, transverse, left, each scored between 0 - 3) and is summed for a total score between 0 - 9.(16, 17)(Appendix A) Adequacy was recently formally defined in a large study involving 2,516 patients undergoing colonoscopies at 36 centres as a total score ≥6 and/or all segment scores ≥2.(18)

The optimal bowel preparation to use for repeat colonoscopy in patients who failed the initial preparation is unknown. However, a combination of a stimulant, such as bisacodyl, and a larger volume of an electrolyte and fluid balanced osmotic laxative, such as PEG, is often used. In a recent case series, Ibanez et al.(19) identified 83 patients with inadequate bowel preparation at their index colonoscopy. 51 patients agreed to a repeat colonoscopy using an 'intensive' regimen consisting of a low fibre diet, bisacodyl, and 3L split dose polyethylene glycol (PEG). Using this regimen, 90% had adequate bowel preparation at the second colonoscopy. However, the bowel preparation at the index colonoscopy was not given in a split dose manner in the majority of patients, which is now the standard of practice due to superior cleansing, and the lack of a control group makes an accurate assessment of efficacy impossible.(1) In another study, patients with inadequate bowel preparation after split dose PEG (4L) were offered a repeat colonoscopy the same day after ingestion of another 2L of PEG or a colonoscopy 1 week later using a low fibre diet, bisacodyl, and 4L split dose PEG.(20) There was no difference in adequacy of bowel preparation although 20% of cases were still inadequate and the lack of randomization and blinding threaten the validity of these results.

To date, no consensus exists regarding the optimal bowel preparation regimen to use in patients with inadequate cleansing due to the absence of clinical trials. Given 4% to 17% of colonoscopies have inadequate bowel preparation, there is a significant public health need to address this issue.(5-12, 21-23) A highly efficacious yet tolerable bowel preparation regimen is needed for these patients to ensure adequate cleansing for their next procedure. The objective of this multi-centre randomized clinical trial will be to compare the efficacy of two regimens in achieving adequate bowel preparation after failing to cleanse at the index colonoscopy.

PROJECT DESCRIPTION

3.1 Study Design, Randomization, and Blinding This multi-centre randomized clinical trial will compare two bowel preparation regimens for patients who have already failed bowel preparation at their index colonoscopy, defined as inadequate visualization to detect lesions > 5 mm and requiring a shortened colonoscopy interval as a result. This clinical definition of failed bowel preparation was chosen instead of the BBPS since the latter may not be available from the index colonoscopy depending on the endoscopist. However, where possible, the BBPS at the index colonoscopy will be recorded. A total of four centres from the original B-CLEAN study group have agreed to participate (Appendix E).

Subjects will be randomized to one of 2 arms (see '3.2 Selection of Bowel Preparation Regimens' for details). Randomization will be performed centrally using Research Electronic Data Capture (REDCap) in a 1:1 allocation in blocks of varying sizes stratified by site. In addition, data entry will be performed online through REDCap.

Blinding of the endoscopist will be strictly enforced. Endoscopists are required to remain blinded to the subject's bowel preparation until after completing the bowel cleanliness section of the CRF. Subjects will be asked to not discuss the bowel preparation with any endoscopy unit staff except for research personnel until the colonoscopy preparation rating has been completed by the endoscopist. Unfortunately, blinding of the patient (ie. double blinding) is impossible due to the volume differences between the two bowel preparation regimens.

3.2 Selection of Bowel Preparation Regimens Regimen A: 4L PegLyte + 15 mg bisacodyl Regimen B: 6L PegLyte + 15 mg bisacodyl

There is no standard bowel preparation utilized after a colonoscopy with failed bowel preparation. Regimen A was adapted from Ibanez et al.(19) who used a regimen consisting of 3L polyethylene glycol (PEG) and 10 mg bisacodyl with reasonable effectiveness. In our study, 4L PEG is used instead of 3L to avoid reducing the amount of PEG consumed by those who were originally prepped with 4L PegLyte at their index colonoscopy. 15 mg bisacodyl was used instead of 10 mg for consistency with dosing used in BiPegLyte. This regimen is modestly more intensive than standard bowel preparation due to an additional 2L PEG compared to BiPegLyte and 15 mg bisacodyl compared to 4L PegLyte.

Regimen B was adapted from Kim et al.(20) as a more intensive yet tolerable regimen. In this regimen, 6L of PEG is combined with 15 mg of bisacodyl.

3.3 Bowel Preparation & Colonoscopy Subjects will be randomized in a 1:1 allocation to either regimen A or B. Regardless of randomization, subjects will be instructed to follow a low fibre diet for 2 days followed by clear fluid diet for 24 hours prior to the scheduled colonoscopy. The time and amount of PEG the subjects will consume will depend on randomization.(APPENDIX B) To optimize patient adherence, all participants will receive a handout with their specific bowel preparation instructions based on their randomization.

All colonoscopies will be performed within 12 weeks of randomization but not within 2 weeks of index colonoscopy (ie. washout period from the index bowel preparation). Procedures will be performed according to local standard operating procedures. All participating endoscopists will complete standardized training and calibration in the use of the Boston Bowel Preparation Scale prior to the start of the study at http://www.bmc.org/gastroenterology/research.htm. A record of training will be sent to the coordinating centre.

For subjects who do not present for their colonoscopy after randomization (ie. forgot appointment), they may remain in the study and be prepped with the same regimen again as long as their next colonoscopy is not scheduled within the next two weeks. For subjects who decline ongoing study participation, they can withdraw and follow up with their physician.

3.4 Baseline Data Collection

1. Age
2. Gender
3. Weight
4. Height
5. Primary Language
6. Highest level of education
7. Patient's ability to understand and follow the bowel preparation directives at home as deemed by the research personnel (Y/N)
8. Charlson co-morbidity index score (24)

7. Irritable bowel syndrome according to ROME III criteria (25) 8. Functional constipation according to ROME III criteria (25) 9. Neurologic disorders: Parkinson's disease, multiple sclerosis, cerebral palsy, other 10. Previous abdominal/pelvic surgery 11. Established diagnosis of inflammatory bowel disease. 12. Medication usage 13. Information regarding index colonoscopy

1. Method of communication for index colonoscopy
2. Bowel preparation used
3. Use of split dose bowel preparation (Y/N)
4. Did patient followed the diet as prescribed (Y/N)
5. Did patient take bowel preparation medication as prescribed (Y/N)
6. Subject willingness to repeat the index bowel preparation
7. Subject incontinence & travel time with index bowel preparation 14. Indication for index colonoscopy (screening, surveillance, diagnostic)

3.5 Statistical Considerations Sample size was calculated as follows. Assuming 70% adequacy among those randomized to regimen A, 87.5% adequacy among those randomized to regimen B, significance of 0.05, and power of 0.8, 85 patients are required in each group (total = 170). An adequacy rate of 70% was selected based on the existing literature.(19, 20) Additional factors considered in arriving at this figure include the lack of split dosing used at the index colonoscopy (19), inadequate intake of PEG at the index colonoscopy (20), and the performance of the second colonoscopy within a week of the first.(20) An adequacy rate of 87.5% was selected based on a 25% relative increase in adequacy to be considered clinically significant. Based on a target sample size of 170 and a conservative 15% dropout, 196 subjects are required for the study.

Descriptive statistics will be reported as mean (SD), median (range), and proportions as appropriate. Data will be analyzed as intention-to-treat and hypothesis testing performed with t-test, chi-square, and Fisher's exact test as appropriate. Pre-planned secondary analyses will include per-protocol analysis, stratification by timing of colonoscopy (ie. morning versus afternoon procedures), and stratification by initial bowel preparation used.

ELIGIBILITY:
Inclusion Criteria:

1. Anyone undergoing a repeat colonoscopy due to failed bowel preparation at index colonoscopy. Failure is defined as preparation quality inadequate to detect lesions > 5 mm after washing and requiring a shortened colonoscopy interval as a result.
2. Age > 18 years
3. Outpatient colonoscopy
4. Indication for full colonoscopy

Exclusion Criteria:

1. Subject refusal
2. Able to comprehend the trial
3. Index colonoscopy performed as an inpatient
4. Pregnancy or breastfeeding
5. Allergies to the employed bowel preparations
6. Any colonic surgery
7. History of ischemic colitis
8. Congestive heart failure
9. Chronic renal failure
10. Cirrhosis
11. Severe electrolyte imbalance
12. Non-adherence to index bowel preparation defined as failure to follow diet instructions and/or consume the entire volume of bowel preparation medication as prescribed for any reason (ex. eating a normal diet on the day of colonoscopy, PEG intolerance, etc…)
13. Use of bowel preparation in an off-label manner for the index colonoscopy.
14. Inability to follow verbal and written instructions in English or French.
15. Ileus, gastric outlet obstruction, gastrointestinal obstruction, bowel preforation
16. Toxic coitis or toxic megacolon
17. Acute surgical abdomen including appendicitis
18. Gastroenteritis and acute diverticulitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation | Once after colonoscopy
  BBPS total score ≥6 and/or all segment scores ≥2.

SECONDARY OUTCOMES:
Mean BBPS total score | Once after colonoscopy
Bowel preparation was adequate after washing to visualize lesions > 5 mm of importance to the procedure and there is no need to shorten the interval of the next colonoscopy | Once after colonoscopy
Validated patient tolerability questionnaire for bowel preparation score | Once after colonoscopy
Bowel preparation related adverse event | After colonoscopy and 14 days after colonoscopy
  The following moderate and non-lasting symptoms related to bowel prep are expected and not considered adverse events:
  * Nausea
  * Vomiting
  * Abdominal fullness
  * Bloating
  * Abdominal cramps and pain
  * Diarrhea
  * Anal irritation
  Otherwise, all AEs will be classified as follows:
  Severity:
  * Mild
  * Moderate
  * Severe
  Causality:
  * Unrelated
  * Possible
  * Probable
  * Highly probable
  Outcome:
  * Resolved without residual effects
  * Resolved with residual effects
  * Recovering/Resolving
  * Not Recovered/Not Resolved
  * Death
  * Unknown
  A Serious Adverse Event (SAE) is defined as an event that
  * Led to a death
  * Led to a serious deterioration in the health of the subject that resulted in a life-threatening illness or injury, permanent impairment of a body structure or function, hospitalization or prolongation of hospitalization, or required medical or surgical intervention to prevent permanent impairment of a body structure or function
Right sided BBPS sub-score | Up to 4 weeks after colonoscopy

OTHER OUTCOMES:
Detection rate by histology (polyp, adenoma, advanced adenoma (>1 cm, villous component, sessile serrated adenoma, or high grade dysplasia), and adenocarcinoma) | Once after colonoscopy
Cecal intubation rate | Once after colonoscopy
Subject product completion (% of total required intake) | Once after colonoscopy
Subject willingness to repeat the preparation | Once after colonoscopy
Subject incontinence & travel time | Once after colonoscopy
Polyp per colonoscopy | Up to 4 weeks after colonoscopy
Adenoma per colonoscopy | Up to 4 weeks after colonoscopy
Fecal incontinence rate | Up to 4 weeks after colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sey, MD, Principal Investigator — Western University
Locations (4):
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - CHUM, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Saltzman JR, Cash BD, Pasha SF, Early DS, Muthusamy VR, Khashab MA, Chathadi KV, Fanelli RD, Chandrasekhara V, Lightdale JR, Fonkalsrud L, Shergill AK, Hwang JH, Decker GA, Jue TL, Sharaf R, Fisher DA, Evans JA, Foley K, Shaukat A, Eloubeidi MA, Faulx AL, Wang A, Acosta RD. Bowel preparation before colonoscopy. Gastrointest Endosc. 2015 Apr;81(4):781-94. doi: 10.1016/j.gie.2014.09.048. Epub 2015 Jan 14. No abstract available. PMID 25595062
- [Background] Rex DK. Optimal bowel preparation--a practical guide for clinicians. Nat Rev Gastroenterol Hepatol. 2014 Jul;11(7):419-25. doi: 10.1038/nrgastro.2014.35. Epub 2014 Apr 1. PMID 24686267
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the U.S. multi-society task force on colorectal cancer. Gastrointest Endosc. 2014 Oct;80(4):543-562. doi: 10.1016/j.gie.2014.08.002. No abstract available. PMID 25220509
- [Background] Yee R, Manoharan S, Hall C, Hayashi A. Optimizing bowel preparation for colonoscopy: what are the predictors of an inadequate preparation? Am J Surg. 2015 May;209(5):787-92; discussion 792. doi: 10.1016/j.amjsurg.2014.12.018. Epub 2015 Feb 12. PMID 25796095
- [Background] MacPhail ME, Hardacker KA, Tiwari A, Vemulapalli KC, Rex DK. Intraprocedural cleansing work during colonoscopy and achievable rates of adequate preparation in an open-access endoscopy unit. Gastrointest Endosc. 2015 Mar;81(3):525-30. doi: 10.1016/j.gie.2014.05.002. Epub 2014 Jul 3. PMID 24998464
- [Background] Dik VK, Moons LM, Huyuk M, van der Schaar P, de Vos Tot Nederveen Cappel WH, Ter Borg PC, Meijssen MA, Ouwendijk RJ, Le Fevre DM, Stouten M, van der Galien O, Hiemstra TJ, Monkelbaan JF, van Oijen MG, Siersema PD; Colonoscopy Quality Initiative. Predicting inadequate bowel preparation for colonoscopy in participants receiving split-dose bowel preparation: development and validation of a prediction score. Gastrointest Endosc. 2015 Mar;81(3):665-72. doi: 10.1016/j.gie.2014.09.066. Epub 2015 Jan 17. PMID 25600879
- [Background] Ben-Horin S, Bar-Meir S, Avidan B. The outcome of a second preparation for colonoscopy after preparation failure in the first procedure. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):626-30. doi: 10.1016/j.gie.2008.08.027. PMID 19251002
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Ness RM, Manam R, Hoen H, Chalasani N. Predictors of inadequate bowel preparation for colonoscopy. Am J Gastroenterol. 2001 Jun;96(6):1797-802. doi: 10.1111/j.1572-0241.2001.03874.x. PMID 11419832
- [Background] Hookey LC, Vanner SJ. Pico-salax plus two-day bisacodyl is superior to pico-salax alone or oral sodium phosphate for colon cleansing before colonoscopy. Am J Gastroenterol. 2009 Mar;104(3):703-9. doi: 10.1038/ajg.2008.167. Epub 2009 Feb 17. PMID 19223885
- [Background] Lebwohl B, Kastrinos F, Glick M, Rosenbaum AJ, Wang T, Neugut AI. The impact of suboptimal bowel preparation on adenoma miss rates and the factors associated with early repeat colonoscopy. Gastrointest Endosc. 2011 Jun;73(6):1207-14. doi: 10.1016/j.gie.2011.01.051. Epub 2011 Apr 8. PMID 21481857
- [Background] Clark BT, Rustagi T, Laine L. What level of bowel prep quality requires early repeat colonoscopy: systematic review and meta-analysis of the impact of preparation quality on adenoma detection rate. Am J Gastroenterol. 2014 Nov;109(11):1714-23; quiz 1724. doi: 10.1038/ajg.2014.232. Epub 2014 Aug 19. PMID 25135006
- [Background] Seeff LC, Richards TB, Shapiro JA, Nadel MR, Manninen DL, Given LS, Dong FB, Winges LD, McKenna MT. How many endoscopies are performed for colorectal cancer screening? Results from CDC's survey of endoscopic capacity. Gastroenterology. 2004 Dec;127(6):1670-7. doi: 10.1053/j.gastro.2004.09.051. PMID 15578503
- [Background] Nationwide Colonoscopy Program for the Uninsured [cited 2015 September 21]. Available from: http://www.colonoscopyassist.com/After_Colonoscopy.html.
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Calderwood AH, Jacobson BC. Comprehensive validation of the Boston Bowel Preparation Scale. Gastrointest Endosc. 2010 Oct;72(4):686-92. doi: 10.1016/j.gie.2010.06.068. PMID 20883845
- [Background] Calderwood AH, Schroy PC 3rd, Lieberman DA, Logan JR, Zurfluh M, Jacobson BC. Boston Bowel Preparation Scale scores provide a standardized definition of adequate for describing bowel cleanliness. Gastrointest Endosc. 2014 Aug;80(2):269-76. doi: 10.1016/j.gie.2014.01.031. Epub 2014 Mar 12. PMID 24629422
- [Background] Ibanez M, Parra-Blanco A, Zaballa P, Jimenez A, Fernandez-Velazquez R, Fernandez-Sordo JO, Gonzalez-Bernardo O, Rodrigo L. Usefulness of an intensive bowel cleansing strategy for repeat colonoscopy after preparation failure. Dis Colon Rectum. 2011 Dec;54(12):1578-84. doi: 10.1097/DCR.0b013e31823434c8. PMID 22067188
- [Background] Kim JW, Han JH, Boo SJ, Ko OB, Park SK, Park SH, Yang DH, Jung KW, Kim KJ, Ye BD, Myung SJ, Yang SK, Kim JH, Byeon JS. Rescue bowel preparation: same day 2 L polyethylene glycol addition, not superior to bisacodyl addition 7 days later. Dig Dis Sci. 2014 Sep;59(9):2215-21. doi: 10.1007/s10620-014-3125-3. Epub 2014 Apr 20. PMID 24748228
- [Background] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Background] Hendry PO, Jenkins JT, Diament RH. The impact of poor bowel preparation on colonoscopy: a prospective single centre study of 10,571 colonoscopies. Colorectal Dis. 2007 Oct;9(8):745-8. doi: 10.1111/j.1463-1318.2007.01220.x. Epub 2007 Mar 7. PMID 17477852
- [Background] Fayad NF, Kahi CJ, Abd El-Jawad KH, Shin AS, Shah S, Lane KA, Imperiale TF. Association between body mass index and quality of split bowel preparation. Clin Gastroenterol Hepatol. 2013 Nov;11(11):1478-85. doi: 10.1016/j.cgh.2013.05.037. Epub 2013 Jun 28. PMID 23811246
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] ASGE Standards of Practice Committee; Pasha SF, Shergill A, Acosta RD, Chandrasekhara V, Chathadi KV, Early D, Evans JA, Fisher D, Fonkalsrud L, Hwang JH, Khashab MA, Lightdale JR, Muthusamy VR, Saltzman JR, Cash BD. The role of endoscopy in the patient with lower GI bleeding. Gastrointest Endosc. 2014 Jun;79(6):875-85. doi: 10.1016/j.gie.2013.10.039. Epub 2014 Apr 2. No abstract available. PMID 24703084
- [Background] Rahimi RS, Singal AG, Cuthbert JA, Rockey DC. Lactulose vs polyethylene glycol 3350--electrolyte solution for treatment of overt hepatic encephalopathy: the HELP randomized clinical trial. JAMA Intern Med. 2014 Nov;174(11):1727-33. doi: 10.1001/jamainternmed.2014.4746. PMID 25243839
- [Derived] Sey MSL, Von Renteln D, Sultanian R, McDonald C, Bouin M, Chande N, Sandhu A, Yan B, Martel M, Barkun A. A Multicenter Randomized Controlled Trial Comparing Two Bowel Cleansing Regimens for Colonoscopy After Failed Bowel Preparation. Clin Gastroenterol Hepatol. 2022 Jun;20(6):e1283-e1291. doi: 10.1016/j.cgh.2021.07.015. Epub 2021 Jul 10. PMID 34256147
- [Derived] Sey MSL, von Renteln D, Sultanian R, McDonald C, Martel M, Barkun A. Multicentre endoscopist-blinded randomised clinical trial to compare two bowel preparations after a colonoscopy with inadequate cleansing: a study protocol. BMJ Open. 2019 Jul 9;9(7):e029573. doi: 10.1136/bmjopen-2019-029573. PMID 31289092